CLINICAL TRIAL: NCT02712710
Title: Does Addition of a Functional Knee Brace Improve Rehabilitation Outcome in Subjects With Osteoarthritis of the Knee?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 20140714R; SKH-8302-104-DR-30 (Other Grant/Funding Number: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2014-11-24; First posted 2016-03-18 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2017-01

CONDITIONS: Knee Osteoarthritis
Keywords: knee, osteoarthritis, brace
MeSH Terms: conditions — Osteoarthritis, Knee; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- wear a functional knee brace (Experimental): 20 subjects with symptomatic medial compartment knee OA, with grade 2 to 4 on Kellgren and Lawrence scale, and showing willing to wear a functional knee brace. All of the subjects received 4 weeks' rehabilitation treatment (3 times a week)
  Interventions: Device: functional knee brace
- no wear a functional knee brace (No Intervention): Another 20 subjects with comparable body height, weight, and sex. All of the subjects received 4 weeks' rehabilitation treatment (3 times a week)

INTERVENTIONS:
Device: functional knee brace — The functional knee brace for OA can decrease abnormal varus torque by external force.
  Arms: wear a functional knee brace

SUMMARY:
The purpose of this study is to investigate the effect of functional knee brace in the subjects with medial compartment knee OA.

DETAILED DESCRIPTION:
20 subjects with symptomatic medial compartment knee OA, with grade 2 to 4 on Kellgren and Lawrence scale, and showing willing to wear a functional knee brace will be recruited into this study. Another 20 subjects with comparable body height, weight, and sex will be served as a control group. All of the subjects received 4 weeks' rehabilitation treatment (3 times a week). VAS pain score, WOMAC index, and SF-36 will be evaluated before the treatment, and 1 month, and 3 months after the start of treatment. Patients' satisfaction will be evaluated at 1 month, and 3 months after start of treatment. Patients' compliance and any adverse events due to wearing of the functional knee brace will also be reported. A 2-by-3, 2-way mixed-model analysis of variance, which had 1 between-subject factor (group: knee brace + PT and PT only) and 1 within subject factor (evaluation time:T0, T1, T2) , was performed. Pair-wise comparisons between groups were performed using an independent t test (if in normal distribution) or Mann-Whitney U test (if not in normal distribution). Investigators hypothesize that addition of a functional knee brace would improve rehabilitation outcome in subjects with knee OA.

ELIGIBILITY:
Inclusion Criteria:

According to the American College of Rheumatology (American College of Rheumatology) diagnosis of unilateral medial knee osteoarthritis, according to Kellgren and Lawrence X-rays are classified as two to four acceptable month rehabilitation therapy, and for the first time dressed Thruster Legacy's functional knee brace. The control group of patients with knee osteoarthritis same conditions, but dressed Thruster Legacy functional knee brace.

Exclusion Criteria:

1. have undergone knee surgery
2. the lateral tibiofemoral joint severe (tibio-femoral joint) disease
3. serious knee ligament laxity
4. knee flexion contracture (flexion contracture) than 20 degrees
5. unable to walk
6. the skin of metal (aluminum) allergy
7. lower extremity vascular lesions or swelling

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2014-10 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2017-10 (Actual)

PRIMARY OUTCOMES:
VAS pain score | 1 month
  To the severity of the pain patients experience pain in itself to make a quantitative expression, assessment methods as follows: a horizontal line 10 cm in length, with zero as the most left office, on behalf of completely pain-free; the far right of the line can imagine the most severe pain, subjects were at rest and walking, according to their degree of sense of pain marked on the straight line. Reliability of this scale up to 0.94.

SECONDARY OUTCOMES:
WOMAC index | 1 month
  Western Ontario McMaster University Osteoarthritis Index (WOMAC Index) is the most commonly used assessment study of knee osteoarthritis by functional scales, including pain, stiffness and function of physical activity and other three items. You can use the record score VAS (visual analog scale) or scale from 0 to 4 five scale. A total of 24 projects, of which pain part 5 projects, while the stiffness and joint function. 2 and 17 projects each. The total score of 100 points, higher scores indicate worse situation. WOMAC for assessing knee osteoarthritis has good reliability and validity.
SF-36 | 1 month
  The SF-36 is a 36-item questionnaire that evaluates the quality of life. It is composed of 8 subscales: physical functioning, role-physical, bodily pain, general health, vitality, social functioning, role-emotional, and mental health. Each subscale has a score range of 0 to 100, with a higher score indicating better health status.Patient's evaluation of the treatment effect. Patient's evaluation of the treatment effect consists of the answer to one question: "Is the treatment effective?" scored on a Likert scale (very effective=1, effective=2, not effective=3, worse=4, much worse=5).

CONTACTS AND LOCATIONS:
Overall Officials: Lin-Fen Hsieh, M.D, Principal Investigator — Shin Kong Wu Ho-Su Memorial Hospital
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

REFERENCES:
- [Derived] Hsieh LF, Lin YT, Wang CP, Liu YF, Tsai CT. Comparison of the effect of Western-made unloading knee brace with physical therapy in Asian patients with medial compartment knee osteoarthritis-A preliminary report. J Formos Med Assoc. 2020 Jan;119(1 Pt 2):319-326. doi: 10.1016/j.jfma.2019.05.024. Epub 2019 Jun 13. PMID 31204145